CLINICAL TRIAL: NCT04146844
Title: Prevalence of Two Major Geriatric Syndromes in Community- Dwelling Older Adults: Sarcopenia and Frailty
Brief Title: Prevalence of Two Major Geriatric Syndromes: Sarcopenia and Frailty
Status: Completed | Type: Observational
Sponsor: Goztepe Training and Research Hospital (Other)
Collaborators: Istanbul Medeniyet University (Other); Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Filiz Demirdağ, Principal Investigator, Umraniye Education and Research Hospital
Other Study IDs: GoztepeTRH1
Record Dates: First submitted 2019-10-28; First posted 2019-10-31 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Sarcopenia; Frailty; Frailty Syndrome
MeSH Terms: conditions — Sarcopenia; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sarcopenia and frailty are two major syndromes in older adults. They are shown to be associated with low levels of functioning and higher rates of morbidity and mortality. In this study, we aim to report the prevalence of sarcopenia and frailty by using simple assessment methods such as SARC-F and FRAIL, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Being at the age of 65 or older

Exclusion Criteria:

* <24 points on Mini-Mental State Examination
* 12 points or higher on Geriatric Depression Scale

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Community-dwelling older adults
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-25 (Actual)

PRIMARY OUTCOMES:
SARC-F | 5 minutes
  SARC-F is a rapid tool to assess sarcopenia in elderly. It is considered indicative sign of sarcopenia if the person scores 4 points or higher out of 10 points.
FRAIL | 5 minutes
  The FRAIL scale (Fatigue, Resistance, Ambulation, Illnesses, & Loss of Weight) is a simple questionnaire of frailty syndrome for older adults. If a patient scores 3-5 points over a total score of 5 points in the FRAIL, he is considered as frail.

SECONDARY OUTCOMES:
Study of Osteoporotic Fracture (SOF) Criteria for Frailty | 5 minutes
  SOF is another index for measuring frailty. 2 or 3 points out of 3 points are considered as cut-off points for frailty.
Charlson Comorbidity Index | 5-10 minutes
  For comorbidity assessment
Rapid Assessment of Physical Activity (RAPA) | 10 minutes
  For the assessment of physical activity level
Mini-Nutritional Assessment (MNA) | 10 minutes
  Assessment of nutritional status
Katz Index of Independence in Activities of Daily Living | 10 minutes
  Assessment of activities of daily living
Lawton -Brody Instrumental Activities of Daily Living Scale | 10 minutes
  Instrumental activities of daily living assessment
Mini-Mental State Examination | 15 minutes
  Mini-Mental State Examination
Blood Sample Analysis | 5 minutes
  A blood sample analysis will be performed to investigate the relationship between blood parameters, sarcopenia and frailty.
Geriatric Depression Scale- Short Form | 10 minutes
  Assessment of depression

CONTACTS AND LOCATIONS:
Locations (1):
- Umraniye Education and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No